CLINICAL TRIAL: NCT01313715
Title: A Phase Ib Clinical Trial for Inactivated Vaccine (Vero Cell) Against EV71 in Chinese Children and Infants
Brief Title: A Clinical Trial for Inactivated Vaccine (Vero Cell) Against EV71 in Chinese Children and Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Bejing Vigoo Biological Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT004
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-03

CONDITIONS: Hand, Foot, and Mouth Disease; Enterovirus Infections
Keywords: Safety; Immunogenicity; inactivated EV71 vaccine
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Enterovirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 160U /0.5ml in children (Experimental): inactivated vaccine(vero cell) against EV71 of 160U /0.5ml in 45 children aged 13-60 months old on day0,28
  Interventions: Biological: 160U /0.5ml
- 320U /0.5ml in children (Experimental): inactivated vaccine(vero cell) against EV71 of 320U /0.5ml in 45 children aged 13-60 months old on day0,28
  Interventions: Biological: 320U /0.5ml
- 640U /0.5ml in children (Experimental): inactivated vaccine(vero cell) against EV71 of 640U /0.5ml in 45 children aged 13-60 months old on day0,28
  Interventions: Biological: 640U /0.5ml
- 160U /0.5ml in infants (Experimental): inactivated vaccine(vero cell) against EV71 of 160U /0.5ml in 45 infants aged 6-12 months old on day0,28
  Interventions: Biological: 160U /0.5ml
- 320U /0.5ml in infants (Experimental): inactivated vaccine(vero cell) against EV71 of 320U /0.5ml in 45 infants aged 6-12 months old on day0,28
  Interventions: Biological: 320U /0.5ml
- 640U /0.5ml in infants (Experimental): inactivated vaccine(vero cell) against EV71 of 640U /0.5ml in 45 infants aged 6-12 months old on day0,28
  Interventions: Biological: 640U /0.5ml
- 0/0.5ml placebo in children (Placebo Comparator): 0/0.5ml placebo in 45 children aged 13-60 months old on day0,28
  Interventions: Biological: 0/0.5ml placebo
- 0/0.5ml placebo in infants (Placebo Comparator): 0/0.5ml placebo in 45 infants aged 6-12 months old on day0,28
  Interventions: Biological: 0/0.5ml placebo

INTERVENTIONS:
Biological: 160U /0.5ml — inactivated vaccine(vero cell) against EV71 of 160U /0.5ml, two doses, one month interval
  Arms: 160U /0.5ml in children; 160U /0.5ml in infants
Biological: 320U /0.5ml — inactivated vaccine(vero cell) against EV71 of 320U /0.5ml, two doses, one month interval
  Arms: 320U /0.5ml in children; 320U /0.5ml in infants
Biological: 640U /0.5ml — inactivated vaccine(vero cell) against EV71 of 640U /0.5ml, two doses, one month interval
  Arms: 640U /0.5ml in children; 640U /0.5ml in infants
Biological: 0/0.5ml placebo — 0/0.5ml placebo, two doses, one month interval
  Arms: 0/0.5ml placebo in children; 0/0.5ml placebo in infants

SUMMARY:
Hand, foot, and mouth disease (HFMD) is a common viral illness in infants and children caused by viruses that belong to the enterovirus genus of the picornavirus family. Although most HFMD cases do not result in serious complications, outbreaks of HFMD caused by enterovirus 71 (EV71) can present with a high rate of neurological complications, including meningoencephalitis, pulmonary complications, and can even cause infant death. HFMD caused by EV71 has become a major emerging infectious disease in Asia and the highly pathogenic potential of EV71 clearly requires the attention of world medical community.

Recently, an inactivated vaccine(vero cell) against EV71 has been licensed by SFDA in China, this clinical trial phase Ib is armed to evaluate safety in Chinese healthy children (from 13 to 60 months old) and infants (from 6 to 12 months old) and also provide the evidences for the EV71 vaccine immunogenicity and the probable immunizing dose.

DETAILED DESCRIPTION:
Hand, foot, and mouth disease (HFMD) is a common viral illness in infants and children caused by viruses that belong to the enterovirus genus of the picornavirus family. Although most HFMD cases do not result in serious complications, outbreaks of HFMD caused by enterovirus 71 (EV71) can present with a high rate of neurological complications, including meningoencephalitis, pulmonary complications, and can even cause infant death. HFMD caused by EV71 has become a major emerging infectious disease in Asia and the highly pathogenic potential of EV71 clearly requires the attention of world medical community.

The development of vaccine against EV71 is active and ongoing in Asian countries now. Several studies have examined the effectiveness of inactivated viral vaccines against EV71 in animal model. A wide range of experimental EV71 vaccine approaches have been studied including heat-inactivated or formaldehyde-inactivated virion, EV71 virus-like particles (VLP) , VP1 recombinant protein ,VP1 DNA vaccine , VP1 peptide-based vaccine targeting the neutralizing domain, bacterial or viral vector expressing VP1, and a Vero cell-adapted live attenuated virus. Furthermore, neutralizing antibodies against EV71 have been suggested as one of the most important factors in prevention of the severe EV71 infection.

Recently, an inactivated vaccine(vero cell) against EV71 has been licensed by SFDA in China, this clinical trial phase Ib is armed to evaluate safety in Chinese healthy children and infants and also provide the evidences for the EV71 vaccine immunogenicity and the probable immunizing dose.

ELIGIBILITY:
For the subjects aged from 13-60 months:

Inclusion Criteria:

* Healthy subjects aged from 13 to 60 months old as established by medical history and clinical examination
* The subjects' guardians are able to understand and sign the informed consent
* Had never received the vaccine against EV71
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature <37.1°C on axillary setting

Exclusion Criteria:

* Subject who has a medical history of HFMD
* <= 37 weeks gestation
* Subjects with a birth weight <2.5 kg
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Severe malnutrition or dysgenopathy
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Autoimmune disease
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6month
* Any prior administration of blood products in last 3 month
* Any prior administration of other research medicines in last 1month
* Any prior administration of attenuated live vaccine in last 28 days
* Any prior administration of inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Under the anti - TB prevention or therapy
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

For the subjects aged from 6-12 months:

Inclusion Criteria:

* Healthy subjects aged from 6 to 12 months old as established by medical history and clinical examination
* The subjects' guardians are able to understand and sign the informed consent
* Had never received the vaccine against EV71
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature <37.1°C on axillary setting

Exclusion Criteria:

* Subject who has a medical history of HFMD
* <= 37 weeks gestation
* Subjects with a birth weight <2.5 kg
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Severe malnutrition or dysgenopathy
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Autoimmune disease
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6month
* Any prior administration of blood products in last 3 month
* Any prior administration of other research medicines in last 1month
* Any prior administration of attenuated live vaccine in last 28 days
* Any prior administration of inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Under the anti - TB prevention or therapy
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events after first vaccination | 28 days after the first vaccination
  To evaluate the adverse events of EV71 vaccine in healthy children and infants after first vaccination
Number of participants with adverse events after second vaccination | 28 days after the second vaccination
  To evaluate the adverse events of EV71 vaccine in healthy children and infants after second vaccination

SECONDARY OUTCOMES:
The seroconversion rate of anti-EV71 antibodies in serum after first vaccination | 28 days after the first vaccination
  To evaluate the seroconversion rate of anti-EV71 antibodies in serum 28 days after first vaccination
The seroconversion rate of anti-EV71 antibodies in serum after second vaccination | 28 days after second vaccination
  To evaluate the seroconversion rate of anti-EV71 antibodies in serum 28 days after second vaccination
The abnormity change of liver and kidney function indexes in serum after first vaccination in children | 3 days after first vaccination
  To evaluate the abnormity change of liver and kidney function indexes in serum 3 days after first vaccination in children
The abnormity change of liver and kidney function indexes in serum after second vaccination in children | 3 days after second vaccination
  To evaluate the abnormity change of liver and kidney function indexes in serum 3 days after second vaccination in children

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Master, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Donghai Center for Diseases Control and Prevention, Lianyungang, Jiangsu, China

REFERENCES:
- [Derived] Mao Q, Cheng T, Zhu F, Li J, Wang Y, Li Y, Gao F, Yang L, Yao X, Shao J, Xia N, Liang Z, Wang J. The cross-neutralizing activity of enterovirus 71 subgenotype c4 vaccines in healthy chinese infants and children. PLoS One. 2013 Nov 19;8(11):e79599. doi: 10.1371/journal.pone.0079599. eCollection 2013. PMID 24260259